CLINICAL TRIAL: NCT01146938
Title: A Clinical Trial to Compare and Evaluate the Pharmacokinetic Characteristics and the Safety of Fimasartan in Hepatic Impairment Patients and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Kyungpook National University Hospital (Other); Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: A657-BR-CT-112
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2010-12

CONDITIONS: Essential Hypertension; Hepatic Impairment
Keywords: fimasartan; hepatic impairment
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hepatic impairment patients (Experimental): Hepatic impairment patients group Child-Pugh score A or Child-Pugh score B (not Child-Pugh score C)
  Interventions: Drug: fimasartan
- Healthy volunteers (Active Comparator): healthy volunteers group
  Interventions: Drug: fimasartan

INTERVENTIONS:
Drug: fimasartan — single administration of fimasartan 120mg
  Arms: hepatic impairment patients
Drug: fimasartan — single administration of fimasartan 120mg
  Arms: Healthy volunteers

SUMMARY:
To compare and evaluate the pharmacokinetic characteristics and the safety of fimasartan in hepatic impairment patients and healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

<Hepatic impairment patient>

* age: 20 - 64 years
* sex: male
* Child-Pugh score A or Child-Pugh score B
* body weight: greater than 55 kg
* written informed consent

<Healthy volunteer>

* age: 20 - 64 years
* sex: male
* body weight: greater than 55 kg
* written informed consent

Exclusion Criteria:

<Hepatic impairment patient>

* portosystemic shunt surgery
* Child-Pugh score C
* creatinine clearance < 80mL/min
* ascites

<Healthy volunteer>

* AST(SGOT), ALT(SGPT) > 1.5 times of Upper Normal Range
* Total bilirubin > 1.5 times of Upper Normal Range
* positive drug or alcohol screening

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic characteristics of fimasartan | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 32, 48h
  AUC, Cmax, Tmax, T1/2, CL/F of fimasartan

CONTACTS AND LOCATIONS:
Overall Officials: Minsoo Park, PhD, Principal Investigator — Yonsei University
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim CO, Lee HW, Oh ES, Seong SJ, Kim DY, Lee J, Ahn SH, Yoon YR, Cho CM, Park MS. Influence of hepatic dysfunction on the pharmacokinetics and safety of fimasartan. J Cardiovasc Pharmacol. 2013 Dec;62(6):524-9. doi: 10.1097/FJC.0000000000000010. PMID 24084213